CLINICAL TRIAL: NCT04095754
Title: Can Anti-Trendelenburg Position Improve Surgical Field Without Affecting Accessibility During Ear Surgery? A Randomized-Controlled Trial.
Brief Title: Can Head Position Improve Surgical Field During Ear Surgery?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hala Salah El-Din El-Ozairy, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: FMASU R 49/2019
Record Dates: First submitted 2019-09-13; First posted 2019-09-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Intra-operative Bleeding
MeSH Terms: interventions — Dexmedetomidine; Hypotension, Controlled; Neoadjuvant Therapy; Anesthetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (control group) (Other): Patients will be positioned supine.
  Interventions: Drug: Dexmedetomidine; Drug: Induction and maintenance of anaesthesia
- Group II (Experimental): patients will be positioned 10° anti-trendelenburg position.
  Interventions: Procedure: Head-Up Position; Drug: Dexmedetomidine; Drug: Induction and maintenance of anaesthesia
- Group III (Experimental): patients will be positioned 20° anti-trendelenburg position.
  Interventions: Procedure: Head-Up Position; Drug: Dexmedetomidine; Drug: Induction and maintenance of anaesthesia

INTERVENTIONS:
Procedure: Head-Up Position — Anti-Trendelenburg Position
  Other Names: Anti-Trendelenburg Position
  Arms: Group II; Group III
Drug: Dexmedetomidine — Controlled hypotension: All patients will receive dexmedetomidine 1mcg. Kg-1 loading dose over 10 min just before induction, followed by continuous infusion of 0.4 mcg.kg-1hr-1
  Other Names: controlled hypotension
Drug: Induction and maintenance of anaesthesia — Induction of anaesthesia: fentanyl 1 μg.Kg-1, propofol 1.5-2 mg.kg -1 titrated to loss of verbal response, atracurium 0.5 mg. Kg-1 to facilitate endotracheal intubation.
  Maintenance:Anaesthesia will be maintained using isoflurane 1 % in oxygen and air mixture 1:1 and atracurium 0.1 mg. Kg-1 every 20 mim.
  Other Names: Anaesthetic drugs

SUMMARY:
Middle ear surgeries utilizes microscope in a narrow field. They are better performed under controlled hypotension, to minimize bleeding and improve surgical field visualization and hence improve results.Head-up or anti-trendelenburg position influences intraoperative bleeding by generating regional ischaemia in sites elevated above the level of the heart. Also by augmenting the effect of vasodilators through pooling of blood in dilated veins.

DETAILED DESCRIPTION:
After obtaining local ethical committee approval and written informed consent from the patients, 225 adult patients, scheduled for elective middle ear surgery in Ain Shams University hospitals will be enrolled in this randomized, prospective controlled study.

After applying basic monitors (ECG, pulse oximetry, non-invasive blood pressure monitoring and capnography), all patients will be premedicated with midazolam 0.02 mg.kg -1 IV and ranitidine 50 mg IV, 15 min. prior to surgery.

All patients will receive dexmedetomidine 1mcg. Kg-1 loading dose over 10 min just before induction, followed by continuous infusion of 0.4 mcg.kg-1hr-1. Rate of infusion will be adjusted to maintain MAP 20% below baseline. Dexmedetomidine infusion will be stopped after graft insertion. Total dexmedetomidine consumption will be recorded.

In the operating room and after 5 min preoxygenation, general anesthesia will be conducted using the same protocol for all patients: fentanyl 1 μg.Kg-1, propofol 1.5-2 mg.kg -1 titrated to loss of verbal response, atracurium 0.5 mg. Kg-1 to facilitate endotracheal intubation.

Anaesthesia will be maintained using isoflurane 1 % in oxygen and air mixture 1:1 and atracurium 0.1 mg. Kg-1 every 20 mim. Positive pressure ventilation will be set to maintain normocapnia.

Patients will be randomly and evenly assigned to one of three groups, 75 patients each.

Group I (control): Patients will be positioned supine. Group II: patients will be positioned 10° anti-trendelenburg position. Group III: patients will be positioned 20° anti-trendelenburg position. Randomization will be done using computer generated list. The anaesthesia nurse recording the data is blinded to the study groups.

At the end of surgery, isoflurane will be discontinued and residual neuromuscular blockade will be reversed. Recovery time will be recorded (Defined as: the time from discontinuation of volatile anaesthetic till the patient is able to respond to verbal command). Patients will then be transferred to PACU.

During surgery, if the surgeon found it difficult to complete the surgery in the anti-trendelenburg (groups II and III), surgery will be continued in the supine position. Patients will still be calculated in the pre-assigned group with recording of such event, and assuming surgeon satisfaction to be 5 in these patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II

Exclusion Criteria:

* Patients with uncontrolled hypertension, coronary artery disease or on beta blockers.
* Cerebrovascular insufficiency.
* Anaemia.
* End stage renal failure.
* Liver cirrhosis.
* Patients with coagulopathy or receiving drugs influencing blood coagulation.
* Pregnancy.
* Known sensitivity to any of the study drugs.
* Patients' refusal to participate in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 225 (Actual)
Dates: Start 2020-04-12 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Quality of surgical field. | Immediately after surgery.
  The surgeon, as well as the surgeon's assistant, will be asked to assess the surgical field using a 5-point scale: 1- no bleeding, 2- minimal bleeding, 3- bleeding easily controlled, 4- bleeding hindering work, 5- bleeding stops work.
Surgical position accessibility. | Immediately after surgery.
  The surgeon satisfaction concerning suitability of patient's position will be evaluated using a 5-point scale: 1- excellent, 2- good, 3- acceptable, 4- bad, 5- very bad.

SECONDARY OUTCOMES:
Total dexmedetomidine consumption. | At the end of surgery
  The total dose of dexmedetomidine used for each patient
Surgical time | At the end of surgery
  duration of surgery (skin to skin time)
Recovery time | At the end of surgery
  the time from discontinuation of volatile anaesthetic till the patient is able to respond to verbal command
Sedation Score | on arrival to the PACU, then every 30 min for the first 2 hours after surgery
  Ramasay sedation score: will be assessed on arrival to the PACU, then every 30 min for the first 2 hours after surgery (1= anxious, agitation or restless; 2= cooperative, oriented, and tranquil; 3= responsive to commands; 4= asleep but with brisk response to light, glabellar tab, or loud auditory stimulus; 5= asleep, sluggish response to glabellar tab, or loud auditory stimulus; 6= asleep, no response).
Analgesia time | first 12 hours after surgery
  time to first rescue analgesic required

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ain Shams University Hospitals, Cairo
  - Ain Shams University, Cairo

IPD SHARING:
Plan to Share IPD: Yes
All primery and secondary outcome data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the publication of the study